CLINICAL TRIAL: NCT02373033
Title: The Effects of a 3-months Dietary Intervention With Folate Enhanced Foods on Folate Status in Healthy Egyptian Women
Brief Title: Folate-Rich Foods Improve Folate Status
Acronym: Folatefood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Swedish University of Agricultural Sciences (Other); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government)
Responsible Party: Principal Investigator, Mohammed Hefni, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Formas Sida Dn 222-2009-1975
Record Dates: First submitted 2015-02-03; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Folic Acid Deficiency
Keywords: Folate; folic acid; intervention trial; folate status; women in childbearing age; food folate
MeSH Terms: conditions — Folic Acid Deficiency | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention: Natural food folate (Active Comparator): Food group consumed folate-rich foods (providing additional 250 μg/d folate).
  Interventions: Other: Natural food folate
- Intervention: Folic acid (Active Comparator): Folic acid group received a folic acid supplement (providing additional 500 μg/d folic acid).
  Interventions: Other: Folic acid
- Intervention: Control (Placebo Comparator): Control group received apple juice containing no folate or folic acid every day.
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Natural food folate — Consumed folate-rich foods (providing additional 250 μg/d folate).
  Other Names: Food folate
  Arms: Intervention: Natural food folate
Other: Folic acid — Received a folic acid supplement (providing additional 500 μg/d folic acid).
  Arms: Intervention: Folic acid
Other: Apple juice — Received apple juice containing no folate or folic acid.
  Arms: Intervention: Control

SUMMARY:
This study evaluates the effects of folate-rich foods regarding improvement of folate status compared with folic acid supplement. A randomized, parallel intervention trial with two active groups (folate-rich foods or folic acid supplement) and one control group (apple juice - 0 µg/d folate) was executed over 12 weeks.

DETAILED DESCRIPTION:
Sixty-two women in reproductive age, apparently healthy, non-smokers, not consuming special diets (vegetarian), not pregnant, not planning conception or not lactating.

A randomized, controlled, parallel intervention trial with two active groups and one blinded control group was carried out for 12 weeks (March to June, 2013). The active food group (n = 21) consumed folate-rich foods (germinated canned faba beans, cookies, orange juice, providing additional 250 μg/d folate); the active folic acid supplement group consumed a supplement (n = 19, providing 500 μg/d folic acid); and the control group (n = 22) received apple juice containing no folate or folic acid) in addition to the freely chosen diet.

Fasted venous blood samples were collected at baseline, two months and three months for quantification of folate in plasma and erythrocytes and of homocysteine in plasma.

ELIGIBILITY:
Inclusion Criteria:

Normal biochemical range for:

* Fasted plasma glucose
* Iron status (haemoglobin, serum ferritin)
* Liver status (aspartate transaminase, alanine transaminase, and γ-glutamyl transferase activities)
* Lipid profile (triglycerides, LDL, HDL)
* Folate status (plasma and erythrocyte folate)
* Plasma total homocysteine (tHcy)
* Vitamin B-12

Exclusion Criteria:

* History of acute or chronic disease
* Use of vitamin or mineral supplements or folic acid fortified foods (within the past one month)
* A body mass index (BMI, in kg/m2) >18 and <30
* Any medication interfering with folate metabolism (e.g., antiepileptic drugs, antibiotics, methotrexate, sulfasalazine, or anticonvulsants), smokers, consuming special diets (vegetarian), pregnancy, planned conception or lactation

Ages: 19 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma folate | (0 and 12 weeks)
  Assessment of plasma folate at baseline, 8 and 12 weeks
Change in erythrocyte folate | (0 and 12 weeks)
  Assessment of erythrocyte folate at baseline, 8 and 12 weeks

SECONDARY OUTCOMES:
Change in plasma total homocysteine | (0 and 12 weeks)
  Assessment of plasma total homocysteine at baseline, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Witthöft, Prof, Principal Investigator — Dept of Food Science, Swedish University of Agricultural Sciences
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Ohrvik VE, Olsson JC, Sundberg BE, Witthoft CM. Effect of 2 pieces of nutritional advice on folate status in Swedish women: a randomized controlled trial. Am J Clin Nutr. 2009 Apr;89(4):1053-8. doi: 10.3945/ajcn.2008.27192. Epub 2009 Feb 3. PMID 19190070